CLINICAL TRIAL: NCT05728593
Title: The Effect of Parent-based Occupational Therapy on Parents of Children With Cerebral Palsy: a Randomised Controlled Trial
Brief Title: The Effect of Parent-based Occupational Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Authors (Unknown)
Responsible Party: Principal Investigator, Gokcen Akyurek, Principle investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA21053
Record Dates: First submitted 2023-01-26; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Palsy; Parents
Keywords: cerebral palsy; coping skills; parents; occupational therapy; stress level
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Researchers were not blinded to group assignments and interventions. However, the participants were blinded about the purpose of the study and the groups they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): Participants (n=15) were randomly selected by the researchers using the coin toss method, and thus the participants were divided into two groups as study (n=8) and control group (n=7) The study group received parent-based occupational therapy, while the control group received standard occupational therapy.
  Interventions: Other: parent-based occupational therapy
- control group (Active Comparator): Participants (n=15) were randomly selected by the researchers using the coin toss method, and thus the participants were divided into two groups as study (n=8) and control group (n=7) The study group received parent-based occupational therapy, while the control group received standard occupational therapy.
  Interventions: Other: Standard occupational therapy intervention

INTERVENTIONS:
Other: parent-based occupational therapy — Parent-based occupational therapy intervention While the therapist, parent and child were in the therapy area in the first session, the child received the same standard occupational intervention as the control group, and during this process, the parents recorded the therapy with a video recorder. In the second 20 minutes, three activities (such as eating, dressing or mobility activities), which had been decided and planned by the parent and the therapist before the session, were performed by the child and helped by the parent and video-recorded by the occupational therapist.
  Arms: study group
Other: Standard occupational therapy intervention — The sessions in this intervention included the creation of a client-based programme to increase each child's individual skills, functions and social participation. Each session lasted 45 minutes and took place twice a week until 10 sessions had been completed.
  Various materials such as toys, blocks, paper and pencils were used to increase the child's participation in daily living, leisure and play activities.
  Arms: control group

SUMMARY:
Background/Aims Parents of children with cerebral palsy face higher levels of stress, anxiety and depression, sadness, exhaustion and burnout. Parent-based therapies have been found to increase parents' satisfaction with therapy, parent-child interactions and reduced parental stress. This study examined the effects of parent-based occupational therapy on stress levels, coping skills, and emotional skills and competencies of parents of children with cerebral palsy.

Methods A total of 15 children and their parents who were admitted to the paediatric rehabilitation unit for occupational therapy were divided into two groups (control group: n=7, study group: n=8) using the coin toss randomisation method. The control group received standard occupational thearpy, while the study group received parent-based occupational therapy for 45 minutes a session, twice a week, until 10 sessions had been completed. Participants were evaluated before and after the intervention.

DETAILED DESCRIPTION:
Cerebral palsy is a disability characterized by movement and posture disorders, loss of motor control, muscle weakness, cognitive deficits, sensory impairment, language and communication problems, and epilepsy, resulting from prenatal, perinatal, and postnatal anomalies. This disability is accompanied by intellectual disability, as well as behavioral and emotional difficulties. Cerebral palsy is one of the main causes of childhood motor disability in developed countries and is reported to affect one out of every 500 births. These effects seen in cerebral palsy have negative consequences regarding social participation. Therefore, interventions for children with cerebral palsy are important and valuable.

Rehabilitation of children with cerebral palsy includes interventions that target the child's problems, skills, opportunities (facilitator), difficulties (obstacle), needs, and relationships with their parents. Occupational therapists plan and apply long-term and follow-up interventions to improve children's independence in their environment, such as self-care, play, school, and leisure time occupations. In studies with children with cerebral palsy, evidence-based interventions, such as constraint-induced movement therapy, hand-arm bimanual intensive training, hand-arm bimanual intensive therapy including lower extremity seem to focus on increasing the functional use of the hemiplegic side.

The Ayres sensory integration intervention approach aims to increase functional skills with necessary sensory experiences and active participation. In addition, the Bobath approach focuses on the child's development at a functional level and being able to participate more in activities by improving muscle tone and postural control. These interventions can be used according to the child's needs. The goal is to improve occupational performance and increase social participation.

The effectiveness of an intervention for children with cerebral palsy is related to the amount and intensity of the treatment, as well as the parent's understanding of their children's skills and ability to interact with their children. Stress, anxiety and depression, sadness, exhaustion, burnout, and disappointment are some of the emotions that negatively affect the interactions of parents with their children, as well as the results of the intervention.

Parent-based intervention approaches include parents in the decision-making and implementation of rehabilitation for their child. Law et al stated that parent-based therapies increased parents' satisfaction with therapy, parent-child interactions and reduced parental stress. Barfoot et al observed that a child with cerebral palsy and his parents achieved both emotional and physical wins through a parent-based intervention.

Novak et al found that parent-based occupational therapy home programs contributed positively to the development of children with cerebral palsy and reduced caregivers' burden. The studies found that the treatment applied to children with cerebral palsy was not sufficient and that parents who spend most of their time at home with their children should be included in the interventions.

It is important to benefit from the parents' expertise and for them to see themselves as a part of the intervention. Therefore the aim of the present study was to examine the effectiveness of the parent-based occupational therapy intervention program on coping skills and stress levels in parents of children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study group, the following inclusion criteria had to be met:

1. Children aged between 3 and 12 years who were diagnosed with cerebral palsy and their parents
2. Willing to participate in the study
3. Able to record videos
4. Having the technological equipment to watch the video.

To be eligible for the study group, the following inclusion criteria had to be met:

1. Children aged between 3 and 12 years who were diagnosed with cerebral palsy and their parents
2. Willing to participate in the study.

Exclusion Criteria:

* 1. Had other neurological and/or psychiatric conditions, such as epilepsy or depression 2. Had a sister or brother with disabilities who attended the centre and received parent-based occupational therapy at the centre where the study was held.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Coping Attitudes Assessment Scale | 6 weeks
  The Coping Attitudes Assessment Scale, designed to measure the ability to cope with problems that may be encountered in daily life, is a 60-question self-report scale scored between 1 and 4 (1: I never do such a thing, 2: I do this a little, 3: I do this moderately, 4: I do this mostly). It has 15 sub-scales. These sub-scales refer to a distinct coping attitude, such as positive reinterpretation and growth, behavioural disengagement, active coping, planning, restrain and denial. A sub-scale with a high score indicates that the individual uses that coping attitude a lot (Carver et al, 1989). The Turkish version has been found to be valid and reliable (Agargün et al, 2005).
Emotional Skills And Competence Questionnaire | 6 weeks
  The Emotional Skills and Competence Questionnaire is used to evaluate emotional skills and competencies. It is a 45-item measurement tool based on a 5-point Likert-type (1: almost never; 5: almost always). It has three sub-scales: perception and understanding, display and naming, and arrangement. A higher score indicates better emotional skills and competence in this sub-scale (Mayer and Salovey, 1997). The Turkish version has been found to be valid and reliable (Vatan, 2015).
Questionnaire on Resources And Stress-F | 6 weeks
  The Questionnaire on Resources and Stress-F was created to evaluate the stress levels in families with children with disabilities. The scale consists of 52 statements that are answered as true or false. It has three sub-scales: dysfunction, pessimism, and parental and family problems (Holroyd, 1987). The Turkish version has been found to be valid and reliable (Kaner, 2002).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No